CLINICAL TRIAL: NCT00295048
Title: Cognitive Remediation for Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); VISN 5 Mental Illness Research, Education and Clinical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: H-24292
Record Dates: First submitted 2006-02-19; First posted 2006-02-22 (Estimated); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Schizophrenia
Keywords: treatment; cognition; schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Computer Assisted Cognitive Remediation (CACR)

SUMMARY:
The purpose of this study is to evaluate the efficacy of an innovative, computer driven cognitive rehabilitation program for individuals with schizophrenia and related disorders.

DETAILED DESCRIPTION:
Schizophrenia is associated with neurocognitive impairment, diminished life satisfaction, lack of independence, and poor functioning in social, occupational and other desired and expected community roles. The personal, social and economic costs of this illness are enormous. Neurocognitive deficits (e.g., slowed thinking, poor attention and memory, inadequate problem solving) are now recognized as core features of the illness, and primary contributors to functional impairment among patients (Bellack, Gold & Buchanan; 1999; Green, 1996). While standard antipsychotic medications improve psychotic symptomatology in many patients, their impact on neurocognition is modest, at best, and dramatic functional deficits remain even after adequate pharmacological treatment (Keefe et al., 1999). Hence, there is growing interest in alternative treatment strategies to address cognitive deficits, including computer-assisted cognitive remediation.

The purpose of this project is to assess the efficacy of a computer-assisted cognitive remediation program we have developed: Computer Assisted Cognitive Remediation (CACR). Fifty individuals with schizophrenia and related disorders will be recruited and randomly assigned to one of two conditions: a) 36 sessions of CACR; or b) 36 sessions of a manualized computer control condition (RC). The efficacy of CACR will be assessed on behavioral performance in three dimensions: (1) on the trained learning exercises, (2) on neuropsychological measures, and (3) on role play based assessments of everyday problem solving. We hypothesize that CACR will be more effective than the control treatment in each domain.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of either schizophrenia or schizoaffective disorder according to DSM-IV criteria
2. Age 18 through 50
3. Subjects will be clinically stable as judged by current outpatient or inpatient treatment staff
4. Primary psychiatric medication is a new generation antipsychotic other than Clozapine and/or a dose of first generation antipsychotic equivalent to 10 mg. of less of haloperidol for one month prior to enrollment.

Exclusion Criteria:

1. Documented history of organic brain disease
2. Documented history of mental retardation
3. Physical limitations (e.g., with hearing or vision) that would interfere substantially with use of computer-based exercises
4. Diagnosis of current Substance Dependence according to DSM-IV criteria
5. Participation in the prior full trial of this remediation program (this exclusion is meant to apply to individuals participating in the full controlled trial, and not to individuals participating in the preliminary sub-study).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2004-11 (Actual); Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
broad cognitive performance (as indexed by a composite of the neuropsychological measures) and on a composite of everyday problem solving

SECONDARY OUTCOMES:
individual cognitive domains and individual everyday problem solving domains, the interaction of treatment with various other variables

CONTACTS AND LOCATIONS:
Overall Officials: Dwight Dickinson, PhD, Principal Investigator — University of Maryland, College Park
Locations (3):
- United States (3):
  - University of Maryland - Walter P. Carter Center, Baltimore, Maryland
  - VA Maryland Health Care Systen, Baltimore, Maryland
  - MOSAIC Community Services, Catonsville, Maryland

REFERENCES:
- [Derived] Dickinson D, Tenhula W, Morris S, Brown C, Peer J, Spencer K, Li L, Gold JM, Bellack AS. A randomized, controlled trial of computer-assisted cognitive remediation for schizophrenia. Am J Psychiatry. 2010 Feb;167(2):170-80. doi: 10.1176/appi.ajp.2009.09020264. Epub 2009 Dec 15. PMID 20008941